CLINICAL TRIAL: NCT06084780
Title: Prospective Case Series of Intestinal and Multivisceral Transplantation for Unresectable Mucinous Carcinoma Peritonei (TRANSCAPE)
Brief Title: Intestinal & Multivisceral Transplantation for Unresectable Mucinous Carcinoma Peritonei (TRANSCAPE)
Acronym: TRANSCAPE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7Z23
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Secondary Malignant Neoplasm of Retroperitoneum; Secondary Malignant Neoplasm of Peritoneum; Pseudomyxoma Peritonei
Keywords: Intestinal Transplantation; Multivisceral Transplantation; Pseudomyxoma Peritonei; Unresectable Mucinous Carcinoma Peritonei; TRANSCAPE
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Alemtuzumab; Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intestinal, Multivisceral or Modified Multivisceral Transplantation (Experimental): Participants will undergo intestinal or modified multivisceral transplantation according to their disease extent. Participants will be followed for 12 months from the day of transplantation. Participants will undergo routine clinical follow-up according to standard protocols for the management of participants after visceral organ transplantation and standard oncological follow-up for participants with PMP.
  Interventions: Procedure: Intestinal, Multivisceral or Modified Multivisceral Transplantation; Drug: Alemtuzumab; Drug: Tacrolimus; Drug: Sirolimus

INTERVENTIONS:
Procedure: Intestinal, Multivisceral or Modified Multivisceral Transplantation — Enrolled participants will enter the active transplant waiting list within one month of signing informed consent for study participation. Participants can be listed for:
  * Isolated small bowel transplant (SBT): transplantation of the donor small intestine
  * Modified multivisceral tran I lant (MMVT): transplantation of the donor pancreas and small intestine, with or without stomach
  * Multivisceral transplant (MVT): transplantation of the donor pancreas, small intestine, and liver, with or without stomach
Drug: Alemtuzumab — A post-transplant, steroid-free immunosuppressive regimen will be utilized and will include Alemtuzumab as Antibody Induction Therapy. Participants will be administered two doses of Alemtuzumab (30 mg IV) on days 0 and 1.
Drug: Tacrolimus — A post-transplant, steroid-free immunosuppressive regimen will be utilized and will include Tacrolimus for maintenance. Participants will have Tacrolimus for the first 3 months. Dosing of Tacrolimus will depend on participant target level, starting with 0.05 mg/Kg bid.
Drug: Sirolimus — A post-transplant, steroid-free immunosuppressive regimen will be utilized and will include Sirolimus for maintenance. Participants will have Sirolimus after 3 months of Tacrolimus. Dosing of Sirolimus will depend on participant target level, starting with 2 mg od.

SUMMARY:
The goal of this prospective phase 2 study is to assess the efficacy and safety of intestinal or multivisceral transplantation for participants with PMP not amenable to other curative-intent treatments. Participants will undergo intestinal/multivisceral transplantation. Participants will be followed for 12 months to assess efficacy and safety.

DETAILED DESCRIPTION:
Pseudomyxoma peritonei (PMP) is a rare clinical entity (approximately 2-4 cases per million people) characterized by extensive dissemination of mucinous ascites in the abdominal cavity. Relentless accumulation of mucin causes progressive abdominal distention, intestinal obstruction, malnutrition, cachexia, and ultimately death. As a rare disease, diagnosis is often late, and usually occurs when the disease is in a clinically advanced stage. The prognosis of PMP has been dramatically improved by the introduction of cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC). While outcomes are favorable for participants with disease amenable to CRS+HIPEC, the therapeutic options for participants with unresectable PMP are limited. Intestinal transplantation represents a therapeutic option in participants with unresectable PMP. Overall survival has been shown to improve with participants with unresectable PMP during an Oxford Transplant Center study. The goal of this study is to corroborate the Oxford results on an American cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed pseudomyxoma peritonei (PMP)

  * Both low-grade mucinous carcinoma peritonei (LMCP) or high-grade mucinous carcinoma (HMCP), with or without signet ring cells as well as primary or recurrent disease, will be eligible.
* PMP disease does not have any extra-abdominal metastases, with the exception of pulmonary involvement (nodal, parenchymal, and pleural).
* PMP disease is extensive and not amenable to operative management, with or without liver, pancreas, stomach, or abdominal wall involvement.

  * Definition of Non-Resectable Disease-

    * Non-resectable PMP disease will be defined as the presence of at least one of the following conditions:

      * 1) Extensive small bowel serosa involvement, where it is not possible to preserve at least 1.5-2 m of small bowel
      * 2) Extensive infiltration of the pancreatic surface
      * 3) Mesenteric involvement causing retraction
      * 4) Need for complete gastric resection
      * 5) Urete1ic obstruction
      * 6) Liver disease with no chance to achieve R0 resection with liver remnant volume > 30%
      * 7) Recurrent disease not amenable to further resection
* Subjects do not have any other available curative treatment options.

  * Subjects can have previous abdominal operations, including CRS+HIPEC.
* Age ≥ 18 and ≤ 75.

  * Pediatric participants were excluded as PMP is a disease that affects adults. Participants > 75 years of age are excluded as they are beyond the commonly accepted transplantability criteria.
* Performance status ECOG ≤ 1.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects with peritoneal carcinomatous originating from an etiology other than PMP.
* Subjects receiving any other investigational agents.
* Subjects with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would either put participation at risk because of participation in the study, may influence the result of the study, or limit compliance with study requirements.
* Pregnant women are excluded from this study because an intestinal transplant is a procedure that is not compatible with a viable pregnancy.
* Subjects who are HIV-positive may be included in the study. HIV testing is required for the study as adequate HIV treatment is required prior to intestinal transplant due to the increased risk of infection following transplantation and treatment with immunosuppressive agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Rate of Survival | 12 months post operative
  To determine overall 12-month survival after intestinal or multivisceral transplantation in participants with unresectable PMP.

SECONDARY OUTCOMES:
Overall Rate of Morbidity | 90 days post operative
  Determine the morbidity of intestinal or multivisceral transplantation for participants with unresectable at 90 days by monitoring severe adverse events as classified according to Clavien-Dindo grade and comprehensive complication index.
Overall Rate of Morbidity | 12 months post operative
  Determine the morbidity of intestinal or multivisceral transplantation for participants with unresectable at 12 months by monitoring severe adverse events as classified according to Clavien-Dindo grade and comprehensive complication index.
Overall Rate of Mortality | 12 months post operative
  Determine cancer-related and transplant-related mortality after intestinal or multivisceral transplantation in participants with unresectable PMP.

CONTACTS AND LOCATIONS:
Overall Officials: Masato Fujiki, MD, PhD, Principal Investigator — Cleveland Clinic Digestive Disease & Surgery Institute (DDSI) , Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Digestive Disease & Surgery Institute (DDSI), Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
As an investigator-initiated protocol, individual participant data will not need to be shared with any other third party. Reported results from this trial will be aggregated data.